CLINICAL TRIAL: NCT04383795
Title: A Prospective Study Analyzing the Change of Gut Microbiome With Antithyroid Drug Treatment of Graves' Disease
Brief Title: Change of Gut Microbiome in the Treatment of Graves' Disease
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Dong Jun Lim, Professor in Division of Endocrinology and Metabolism, Department of Internal Medicine, Seoul St. Mary's Hospital, Seoul St. Mary's Hospital
Other Study IDs: KC19TESI0523
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Graves' Disease
MeSH Terms: conditions — Graves Disease | interventions — Antithyroid Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool sample from study participants before and after 6-month antithyroid drug treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Graves' disease patients: First diagnosed Graves' disease patients volunteered for stool collection
  Interventions: Drug: Antithyroid Drug

INTERVENTIONS:
Drug: Antithyroid Drug — Administration of antithyroid Drug for 6 months

SUMMARY:
Graves' disease is the main cause of hyperthyroidism. Graves' disease has a prevalence of 0.5% in the general population. As a non-surgical treatment, antithyroid drug (ATD) and radioactive iodine treatment have been proposed and ATD is the first-line treatment in Korea. However, ATD has a rare but fatal side effect of agranulocytosis. Furthermore only half of its users maintain long-term remission and frequent recurrence is a problem to this disease. Therefore it is essential to distinguish between patients who respond well to ATD and those who resist it. The aim of this study is to verify the changes in gut microbiome in Graves' disease patients before and after six-month treatment with ATD. Patients first diagnosed with Graves' disease will participate in the study. The study design is a prospective longitudinal trial. The patients are asked to have their gut microbiome analyzed before and after the treatment of Graves' disease with ATD. Primary endpoint is the changes of analyzed gut microbiome before and after ATD treatment. Secondary outcome is to find species that can be used as a biomarker to differentiate the patients refractory to ATD.

ELIGIBILITY:
Inclusion Criteria:

* More than 19 years and lesser than 70 years
* First diagnosed as Graves' disease and planned to have antithyroid drug

Exclusion Criteria:

* Pregnancy and lactating women
* Inflammatory bowel disease
* Active malignancy
* Autoimmune disease
* Immune-deficiency patients

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients first diagnosed with Graves' disease, aged more than 19 years and lesser than 70 years. Eligible for treatment of graves' disease with antithyroid drug. Consented for collection of stools in 6-month interval
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change of gut microbiome in the treatment of Graves' disease | 6 months after treatment
  Analysis of gut microbiome before and after treatment of Graves' disease with antithyroid drug

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Jun Lim, MD, PhD, Principal Investigator — the Catholic Univerisity of Korea
Locations (1):
- Seoul St. Mary hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided